CLINICAL TRIAL: NCT06184906
Title: Preventing Celiac Disease by Weaning With Mediterranean Diet
Acronym: PEMED
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Naples (Other)
Responsible Party: Principal Investigator, Luigi Greco, Professor of Pediatrics, University of Naples
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PREVENTCELIAC
Record Dates: First submitted 2023-11-23; First posted 2023-12-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Weaning Failure
Keywords: Infant Weaning; Mediterranean Diet; Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: FP will be randomly assigned in a parallel 1:1 fashion to one of two intervention groups. A block randomization procedure will be considered for the allocation of FP to the intervention. To ensure unbiased allocation, this sequence will be concealed from investigators. Investigative sites will access the randomization information of enrolled participants through a dedicated online system via the RedCap interface10. In line with ethical considerations, enrolled participants and investigators will not be blinded to the study treatments, as the nature of the dietary intervention does not permit blinding. Therefore, unblinding will not be applicable in this trial. As part of the consent process, participants' permission will be sought to use their data even if they choose to withdraw from the trial. Additionally, participants will be asked for consent to share relevant data with researchers from participating universities or regulatory authorities, where relevant.
Who Masked: Outcomes Assessor
Masking Description: Data manager are blind to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROLS (Placebo Comparator): Participants in the control arm will undergo a traditional weaning process. This involves primarily the use of industrial baby foods, with a gradual introduction of fresh foods. Legumes will be introduced at around 7-8 months, and fresh fish will be incorporated into the diet after one year of age.
  Interventions: Dietary Supplement: Weaning by Mediterranean Diet
- Treated (Experimental): Participants in the experimental arm will follow a Mediterranean Diet (MD) weaning schema. This approach includes exclusively fresh foods that are part of the traditional MD, modified to suit infants. Key elements of this diet include:
  * Seasonal fruit and vegetables, such as broccoli and cauliflower, served as purees from the beginning of weaning.
  * A variety of fresh blue fish (e.g., anchovies, mackerel, flag fish, cod, sole) introduced at 7 months, seasoned with garlic and cherry tomatoes.
  * Use of spices and herbs like thyme, marjoram, rosemary, parsley, garlic, and onion to flavor meals.
  * Exclusion of salt; meals are instead enhanced with 2 g of Parmesan cheese for taste.
  * Avoidance of sweets.
  Interventions: Dietary Supplement: Weaning by Mediterranean Diet

INTERVENTIONS:
Dietary Supplement: Weaning by Mediterranean Diet — Introduce solid foods typical of the Mediterranean Diet at weaning of infants

SUMMARY:
Background: The introduction of solid foods in alignment with the Mediterranean Diet (MD) post-exclusive milk feeding has been demonstrated to cultivate a lasting affinity for healthy eating during infancy and childhood. Despite this, access to healthy diets remains a challenge for numerous children, particularly in underserved areas. The clinical trial under discussion is set in Scampia, a municipality in Naples, Italy, known for its dense population and socio-economic challenges. This trial, utilizing the Family Pediatrician (FP) system, aims to promote MD nutrition among children in Scampia to potentially prevent or reduce chronic childhood diseases.

Study Design: In this pragmatic trial, FPs are utilized as the unit for randomization to administer the intervention. The intervention group will be introduced to an intensified MD-based diet from weaning, incorporating adult-type MD foods, while the control group will follow standard regional dietary guidelines. Dietary adherence and health outcomes are to be periodically monitored, and genetic and microbiome analyses will be conducted using collected saliva and stool samples. Incorporating a Bayesian group sequential design, this trial is structured to conduct interim analyses for efficacy, aligning with local healthcare systems for optimal resource allocation.

Conclusion: The study is poised to be methodologically innovative and socially impactful, utilizing existing healthcare frameworks to enhance childhood nutrition in challenging environments. Outcomes from this trial are expected to provide valuable insights into the effects of MD-based nutrition on child health and potentially serve as a model for promoting healthier diets in urban suburbs globally.

DETAILED DESCRIPTION:
Detailed Description:

The relationship between systemic chronic inflammation and various chronic diseases, such as obesity, diabetes, cancer, autoimmune, and inflammatory bowel diseases, is well-recognized. Given the economic impact of these diseases on healthcare systems, a comprehensive strategy for risk prevention is imperative. Diet and intestinal dysbiosis are identified as major triggers for systemic chronic inflammation. The MD, characterized by its anti-inflammatory qualities, has also been noted for its positive effects on gut microbiota. The timing of introducing the MD is critical for fostering a healthy microbiota, with early exposure being advantageous. Furthermore, early dietary experiences are crucial in shaping future food preferences. Evidence suggests that responsive feeding practices, such as baby-led weaning, may offer protection against obesity. While the early introduction of the MD in children remains under-researched, its potential protective role against diseases like celiac and inflammatory bowel diseases has been suggested. The PEMED trial, designed to promote MD nutrition among children in Scampia, represents a groundbreaking approach, utilizing a Bayesian cluster randomized clinical trial and the Italian family pediatrician system.

This study is unique in its exploration of introducing natural MD foods during infancy and assessing their impact on the establishment of lasting dietary preferences. It leverages the healthcare infrastructure of the Piscinola-Scampia district in Naples for a population-based Pragmatic Clinical Trial, exceeding traditional research design norms. The study is focused on assessing the impact of the MD on the incidence of diseases, employing a Bayesian adaptive sequential approach to allow for ongoing data analysis and adjustments. The PEMED trial's novel approach, combining the early introduction of the MD, population-based surveillance, and an advanced statistical methodology, is poised to set new benchmarks in pediatric research concerning diet and disease prevention.

The trial's objectives include evaluating the impact of the MD on the incidence of pediatric diseases, assessing the development of a 'protective' fecal microbiome, and analyzing the persistence of MD dietary choices in children up to the age of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* - Healthy newborns with a birth weight greater than 2000 grams.
* Residence in Municipality 8, Piscinola-Scampia.

Exclusion Criteria:

* - Newborns suffering from severe prematurity.
* Newborns with congenital malformations.
* Newborns afflicted by severe diseases.

Ages: 1 Month to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3200 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Celiac Disease | 3 to 6 years of age
  Monitoring the incidence of Celiac Disease in the study population.
Children growth | 4 to 6 years
  Calculating the Body Mass Index (BMI kg/m^2) as a measure of growth, assessing if children's BMI falls within the normal range for their age and sex.

SECONDARY OUTCOMES:
Beneficial Microbiome | 5 to 6 years of age
  Evaluating the composition of the microbiome for beneficial characteristics.
Bifidibacteriaceae in the feces | 5 years
  Measuring the variation of Bifidobacteria in feces.

IPD SHARING:
Plan to Share IPD: No